CLINICAL TRIAL: NCT06963255
Title: Résultats Des Allogreffes artérielles conservée à +2/+8°C Dans Les REvascularisations en MIlieu Septique
Brief Title: Outcomes of Arterial Allografts Preserved at +2 to +8°C for Revascularization in Septic Settings
Acronym: AREMIS
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5415
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Revascularization in a Septic or Potentially Septic Environment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- The study group will include all patients requiring bypass revascularization in a septic or high-ris: The study group will include all patients requiring bypass revascularization in a septic or high-risk septic environment, for whom a biomaterial is preferred over a prosthetic graft due to the unavailability of the patient's autologous saphenous vein
  Interventions: Procedure: arterial revascularization

INTERVENTIONS:
Procedure: arterial revascularization — arterial revascularization

SUMMARY:
This study does not modify patient management or treatment. All patients undergoing treatment with an arterial allograft preserved at +2/+8°C as part of an arterial revascularization in a septic environment in either of the two centers between January 2024 and January 2025 will be included.

Imaging exams and clinical follow-up data will be analyzed. Reinterventions and causes of death will be recorded. All imaging required for the 6-month follow-up is routinely performed as part of standard care. No modification of patient management is planned.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Requiring revascularization in a septic or high-risk septic environment
* With an estimated life expectancy of 12 months or more based on medical and surgical assessment
* Informed about the study

Exclusion Criteria:

* Pregnant women
* Individuals for whom regular medical follow-up cannot be ensured

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population includes all patients requiring bypass revascularization in a septic or high-risk septic environment, for whom a biomaterial is preferred over a prosthetic graft due to the unavailability of the patient's autologous saphenous vein
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the 6-month primary patency of revascularizations using arterial allografts preserved at +2 to +8°C | 6 month
  Evaluation of the 6-month primary patency of the revascularization, defined as the percentage of patients with a patent bypass without reintervention or >50% stenosis, confirmed by a morphological imaging exam (Doppler ultrasound or CT angiography) performed at 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux
  - HCL hopital Louis Pradel, Bron